CLINICAL TRIAL: NCT00235170
Title: ARTS II: Arterial Revascularization Therapies Study Part II of the Sirolimus-Eluting Bx VELOCITY™ Balloon Expandable Stent in the Treatment of Patients With de Novo Coronary Artery Lesions.
Brief Title: The Arterial Revascularization Therapies Study Part II.
Acronym: ARTS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC01-03
Record Dates: First submitted 2005-10-04; First posted 2005-10-10 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cypher Sirolimus-eluting Coronary stent
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug-eluting stent — Cypher Sirolimus-eluting Coronary stent

SUMMARY:
The main objective is to compare the effectiveness of coronary stent implantation using the sirolimus-eluting Bx VELOCITY™ balloon expandable stent with that of surgery as observed in ARTS I. Effectiveness is measured in terms of Major Cardiac and Cerebrovascular Events (MACCE) free survival at 1 year.

DETAILED DESCRIPTION:
ARTS II is a multicenter, European, open-label, non-randomized, stratified trial in about 45-50 centers which will include six hundred eligible patients with multivessel disease who should be equally treatable by surgery or stenting. In all patients the sirolimus-eluting Bx VELOCITY™ balloon expandable stent of Cordis will be used for treatment.The results of ARTS II will be compared with the by-pass arm of ARTS I as the historical control. It is hypothesized that a similar or higher number of lesions will be treated by stenting. We assume that the use of this eluting stent will not only reduce the rate of MACCE at 30 days, but that it will considerably reduce the need for re-intervention, which was historically 21.0% in ARTS I.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable (Canadian Cardiovascular Society 1, 2, 3 or 4) or unstable (Braunwald class IB, IC, IIB, IIC, IIIB, IIIC) angina pectoris and ischemia, or patients with atypical chest pain or even those who are asymptomatic provided they have documented myocardial ischaemia (e.g. treadmill exercise test, radionuclide scintigraphy, stress echocardiography, Holter tape);
2. Patients who are eligible for coronary revascularization (angioplasty or CABG);
3. At least 2 lesions (located in different vessels and in different territories) potentially amenable to stent implantation;
4. de novo native vessels;
5. Multivessel disease with at least one significant stenosis in LAD and with treatment of the lesion in another major epicardial coronary artery. A two-vessel disease or a three-vessel disease may be viewed as a combination of a side branch and a main epicardial vessel provided they supply different territories; left anterior descending, left circumflex and right coronary artery);
6. Total occluded vessels. One total occluded major epicardial vessel or side branch can be included and targeted as long as one other major vessel has a significant stenosis amenable for SA, provided the age of occlusion is less than one month e.g. recent instability, infarction with ECG changes in the area subtended by the occluded vessel. Patients with total occluded vessels of unknown duration or existing longer than one month and a reference over 1.50 mm should not be included, not even as a third or fourth vessel to be dilated;
7. Significant stenosis has been defined as a stenosis of more than 50% in luminal diameter (in at least one view, on visual interpretation or preferably by QCA);
8. Left ventricular ejection fraction should be at least 30%.

Exclusion Criteria:

1. Congestive heart failure;
2. CABG or Percutaneous Coronary Intervention (PCI) procedure;
3. Planned need for major surgery (e.g. valve surgery or resection of aortic or left ventricular aneurysm, carotid end-arterectomy, abdominal aortic aneurysm surgery etc.);
4. Congenital heart disease;
5. Transmural myocardial infarction within the previous seven days and CK has not returned to normal;
6. Chest pain lasting longer than 30 minutes within 12 hours pre-procedure, if CK enzymes positive (≥ 2x the normal upper limit).
7. History of any cerebrovascular accident;
8. Left main stenosis of 50% or more;
9. Intention to treat more than 1 totally occluded major epicardial vessel;
10. Single vessel (single territory) disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2003-02; Primary Completion 2004-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
abscence of major adverse cardiac and cerebral vascular events (MACCE) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W. Serruys, MD, PhD, Principal Investigator — Thoraxcenter, Erasmus Medical Center, Rotterdam
Locations (1):
- Thoraxcenter, Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Result] Tsuchida K, Colombo A, Lefevre T, Oldroyd KG, Guetta V, Guagliumi G, von Scheidt W, Ruzyllo W, Hamm CW, Bressers M, Stoll HP, Wittebols K, Donohoe DJ, Serruys PW. The clinical outcome of percutaneous treatment of bifurcation lesions in multivessel coronary artery disease with the sirolimus-eluting stent: insights from the Arterial Revascularization Therapies Study part II (ARTS II). Eur Heart J. 2007 Feb;28(4):433-42. doi: 10.1093/eurheartj/ehl539. Epub 2007 Jan 31. PMID 17267457
- [Result] Valgimigli M, Dawkins K, Macaya C, de Bruyne B, Teiger E, Fajadet J, Gert R, De Servi S, Ramondo A, Wittebols K, Stoll HP, Rademaker TA, Serruys PW. Impact of stable versus unstable coronary artery disease on 1-year outcome in elective patients undergoing multivessel revascularization with sirolimus-eluting stents: a subanalysis of the ARTS II trial. J Am Coll Cardiol. 2007 Jan 30;49(4):431-41. doi: 10.1016/j.jacc.2006.06.081. Epub 2007 Jan 12. PMID 17258088
- [Result] Khattab AA, Daemen J, Richardt G, Rioux P, Amann FW, Levy R, Horvath IG, Teles RC, Ordoubadi F, Pieters M, Wittebols K, Stoll HP, Serruys PW. Impact of body mass index on the one-year clinical outcome of patients undergoing multivessel revascularization with sirolimus-eluting stents (from the Arterial Revascularization Therapies Study Part II). Am J Cardiol. 2008 Jun 1;101(11):1550-9. doi: 10.1016/j.amjcard.2008.02.034. Epub 2008 Apr 9. PMID 18489932
- [Result] Daemen J, Kuck KH, Macaya C, LeGrand V, Vrolix M, Carrie D, Sheiban I, Suttorp MJ, Vranckx P, Rademaker T, Goedhart D, Schuijer M, Wittebols K, Macours N, Stoll HP, Serruys PW; ARTS-II Investigators. Multivessel coronary revascularization in patients with and without diabetes mellitus: 3-year follow-up of the ARTS-II (Arterial Revascularization Therapies Study-Part II) trial. J Am Coll Cardiol. 2008 Dec 9;52(24):1957-67. doi: 10.1016/j.jacc.2008.09.010. PMID 19055986
- [Result] Kukreja N, Serruys PW, De Bruyne B, Colombo A, Macaya C, Richardt G, Fajadet J, Hamm C, Goedhart D, Macours N, Stoll HP; ARTS-II Investigators. Sirolimus-eluting stents, bare metal stents or coronary artery bypass grafting for patients with multivessel disease including involvement of the proximal left anterior descending artery: analysis of the Arterial Revascularization Therapies study part 2 (ARTS-II). Heart. 2009 Jul;95(13):1061-6. doi: 10.1136/hrt.2008.157735. Epub 2009 Mar 19. PMID 19304671
- [Derived] Garg S, Sarno G, Garcia-Garcia HM, Girasis C, Wykrzykowska J, Dawkins KD, Serruys PW; ARTS-II Investigators. A new tool for the risk stratification of patients with complex coronary artery disease: the Clinical SYNTAX Score. Circ Cardiovasc Interv. 2010 Aug;3(4):317-26. doi: 10.1161/CIRCINTERVENTIONS.109.914051. Epub 2010 Jul 20. PMID 20647561